CLINICAL TRIAL: NCT00264823
Title: Nursing Intervention for HIV Regimen Adherence Among Serious Mental Illness (SMI)
Brief Title: Nursing Intervention for HIV Regime Adherence Among People With Serious Mental Illness (SMI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Michael B. Blank, PhD, Center for Mental Health Policy and Services Research Department of Psychiatry University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 708134; 5R01NR008851-03 (NIH)
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: HIV; Mental Illness
Keywords: HIV; Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Experimental (Experimental)
  Interventions: Behavioral: Use of Memory Aids to take medications
- 2 - Control (No Intervention)

INTERVENTIONS:
Behavioral: Use of Memory Aids to take medications — Experimental participants will receive an integrated intervention tailored to the communication and comprehension of the individual, and will include memory aid devices, education regarding side effects and other treatment aspects, and active community outreach. For those who fail to adhere using the basic intervention, a treatment cascade that increases in intensity will be implemented. Using 80% adherence as a target, the cascade will include involvement of family and significant others in prompting participants through use of beepers, cellphones, and for those who still fall short of 80% adherence, directly observed therapy.
  Arms: 1 - Experimental

SUMMARY:
The purpose of this research study is to investigate how nurses can best help people with serious mental illnesses (SMI) follow their HIV treatment plans.

DETAILED DESCRIPTION:
There is concern that HIV positive SMI persons may be a greater risk for poor treatment adherence, increasing risk for poorer outcomes and development of treatment resistance virus, and also placing others at greater risk. Involvement of advance practice nurses has been previously shown to improve outcomes for persons with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of serious mental illness; HIV positive

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
How to best help people with serious mental illness follow HIV treatment regimens | baseline, 3, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blank, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Mental Health Services and Policy Research, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Dalseth N, Reed RS, Hennessy M, Eisenberg MM, Blank MB. Does Diagnosis Make a Difference? Estimating the Impact of an HIV Medication Adherence Intervention for Persons with Serious Mental Illness. AIDS Behav. 2018 Jan;22(1):265-275. doi: 10.1007/s10461-017-1795-5. PMID 28536741
- [Derived] Wu ES, Rothbard A, Holtgrave DR, Blank MB. Determining the Cost-Savings Threshold for HIV Adherence Intervention Studies for Persons with Serious Mental Illness and HIV. Community Ment Health J. 2016 May;52(4):439-45. doi: 10.1007/s10597-014-9788-6. Epub 2014 Dec 23. PMID 25535041
- [Derived] Blank MB, Hennessy M, Eisenberg MM. Increasing quality of life and reducing HIV burden: the PATH+ intervention. AIDS Behav. 2014 Apr;18(4):716-25. doi: 10.1007/s10461-013-0606-x. PMID 24000053